CLINICAL TRIAL: NCT04647175
Title: Aronia in the Type 2 Diabetes Treatment Regimen
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1-10-72-102-19
Record Dates: First submitted 2020-11-20; First posted 2020-11-30 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Aronia
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Fermented aronia - aronia - placebo (Other): The participants receive each intervention for 8 weeks in the stated order.
  Interventions: Other: Fermented aronia; Other: Aronia; Other: Placebo
- Fermented aronia - placebo - aronia (Other): The participants receive each intervention for 8 weeks in the stated order.
  Interventions: Other: Fermented aronia; Other: Aronia; Other: Placebo
- Placebo - aronia - fermented aronia (Other): The participants receive each intervention for 8 weeks in the stated order.
  Interventions: Other: Fermented aronia; Other: Aronia; Other: Placebo
- Placebo - fermented aronia - aronia (Other): The participants receive each intervention for 8 weeks in the stated order.
  Interventions: Other: Fermented aronia; Other: Aronia; Other: Placebo
- Aronia - placebo - fermented aronia (Other): The participants receive each intervention for 8 weeks in the stated order.
  Interventions: Other: Fermented aronia; Other: Aronia; Other: Placebo
- Aronia - fermented aronia - placebo (Other): The participants receive each intervention for 8 weeks in the stated order.
  Interventions: Other: Fermented aronia; Other: Aronia; Other: Placebo

INTERVENTIONS:
Other: Fermented aronia — Given twice daily for 8 weeks
Other: Aronia — Given twice daily for 8 weeks
Other: Placebo — Given twice daily for 8 weeks

SUMMARY:
In a triple-crossover study, the effect aronia consumption on type 2 diabetes will be examined. 48 type 2 diabetes patients need to complete the trial. Each patient will receive two daily doses of both fermented aronia, aronia, or placebo for eight weeks each. There will be 3 weeks wash-out periods between the intervention periods. Before and after the intervention periods, various measurements will be performed to assess the effects of aronia, fermented aronia, and placebo on type 2 diabetes.

DETAILED DESCRIPTION:
Hypothesis: Fermented aronia extract (FAE) improves glycaemia and lipidaemia in T2D more efficiently than both non-fermented aronia extract (NFAE) and placebo.

Research questions:

Does FAE/NFAE when administered to T2D subjects:

* Improve glucose responses to an oral glucose tolerance test and HbA1C?
* Improve fasting LDL-, HDL- and total cholesterol?
* Reduce insulin resistance and increase total antioxidative/anti-inflammatory capacity?
* Increase circulating GLP-1 and GIP levels with lower DPP4 activity?
* Alleviate hypertension and obesity?

Methods A total of 48 T2D patients is needed for the double blind, randomized triple cross-over trial. The patients will consume FAE, NFAE or placebo daily divided into two doses which is expected to provide a sufficient dose of bioactive phenolic compounds. The patients will be recruited through "forsoegsperson.dk", "sundhed.dk", and flyers placed at Aarhus university hospital (AUH). T2D patients with fasting blood glucose ≤ 12 mM and HbA1c > 6.1% and < 10%, without severe comorbidities, will be included. Before enrolment, the patients receive all necessary study information (written and oral) including potential adverse effects (e.g. aronia allergy), and they will have to provide their informed consent (visit 1). There will be an assessment of whether the patients fulfill the criteria as well.

The randomized double-blinded triple cross-over study consists of three eight weeks intervention periods (placebo, FAE and NFAE), where the participants are randomly assigned to the order of treatments (six different possibilities of order). The intervention periods are separated by minimum three weeks wash-out periods (see figure 1 for details). Before and after each intervention period, i.e. six times, oral glucose tolerance tests (OGTT) will be performed. The Central Denmark Region Committees on Health Research Ethics has approved the trial.

Analyses OGTT: Prior to the OGTT, the participants have fasted for 8 hours where after they will consume 75 g glucose dissolved in 300 ml water within 5 minutes. Blood will be sampled at time points -10, 0, 30, 60, 90, 120, and 240 minutes.

Blood Analyses: After the blood sampling, plasma will be stored at -80° C until further analysis. Obviously, the investigators aim to determine if FAE and NFAE consumption is capable of lowering the fasting and postprandial blood sugar and thus, the levels of glucose, fructosamin and HbA1c will be measured. The concentration of advanced glycosylation end products will be assessed in fasted blood samples. Also, lipidaemia will be examined, e.g. total cholesterol, triglyceride, high-density lipoprotein and low-density lipoprotein concentrations. The inflammatory state will be assessed by measuring the level of pro- and anti-inflammatory cytokines as well as the concentration of C-reactive protein in fasting blood samples. To determine whether aronia acts through incretin mediated regulation, the concentrations of GIP and GLP-1 and the activity of DDP4 will be measured. The concentrations of glucagon, insulin, and adiponectin will be assessed as well.

Insulin resistance: β-cell dysfunction and insulin resistance will be estimated from blood glucose and insulin concentrations using Homeostasis Model Assessment (3) and Matsuda Index (4) which are based on concentrations measured at fasting states and during the OGTT, respectively.

Diurnal blood pressure: 24-hour ambulatory blood pressure monitoring will be carried out. The necessary equipment is available at AUH. The participants will have their 24-hour blood pressure measured before and after each intervention period.

Body mass index (BMI): At the first visit the participants height and weight are measured, and the weight will subsequently be monitored.

Metabolomics and microbiomics assays: The results from the previous tests (effects on main outcomes) will determine the extent of the subsequent metabolomics and microbiomics analyses. Fecal samples for microbiomics, as well as blood and urine samples for metabolomics will be stored at -80° C until use.

Data analysis: The power calculation is based on our primary effect parameter glucose incremental area under the curve (iAUC). The number of participants needed to obtain a statistical power of 80% at a level of P<0.05 (α=0.05; 1-β=0.8) was calculated as 48. The investigators wanted to detect a minimal relevant difference for the area of (mean ± s.d.) 65±50 mmol/l x 120 min, which gives us an estimated effect size of 1.30. The anticipated dropout is 20%. ANOVA will be conducted for each variable to determine if the variables change upon administration of FAE, NFAE, or placebo as well as to assess intergroup variability at baseline and endpoint. Significance will be set to p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* ≥30 ≤80 years of age
* Fasting blood glucose ≤12 mmol/liter.
* HbA1c > 6,1% og <10%(>43 og < 86 mmol/mol) if patients are in medical diabetes treatment
* HbA1c > 6,5% og <10% (>48 og < 86 mmol/mol) if patients are not in medical diabetes treatment

Exclusion Criteria:

* Changes in diabetes within the last 3 months.
* Serious comorbidities, including cardiovascular-, neurological-, psychological- and/or renal diseases.
* Pregnant or planned pregnancy.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2020-11-23 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Blood glucose incremental area under the curve (iAUC) | Throughout the study (up to 1 year)
  Measured during the OGTTs
Blood glucose total area under the curve (tAUC) | Throughout the study (up to 1 year)
  Measured during the OGTTs

SECONDARY OUTCOMES:
Glucose | Throughout the study (up to 1 year)
  Measured in blood and urin, fasting + during OGTT
Insulin | Throughout the study (up to 1 year)
  Measured in blood, fasting + during OGTT
HbA1c | Throughout the study (up to 1 year)
  Measured in blood, fasting
Fructosamin | Throughout the study (up to 1 year)
  Measured in blood, fasting
Lipids | Throughout the study (up to 1 year)
  Measured in blood, fasting
C-reactive protein | Throughout the study (up to 1 year)
  Measured in blood, fasting
Adiponectin | Throughout the study (up to 1 year)
  Measured in blood, fasting
Inflammatory and oxidative markers | Throughout the study (up to 1 year)
  Measured in blood, fasting
Incretins | Throughout the study (up to 1 year)
  Measured in blood, fasting
DPP4 activity | Throughout the study (up to 1 year)
  Measured in blood, fasting
Advanced glycation end products | Throughout the study (up to 1 year)
  Measured in blood, fasting
Glucagon | Throughout the study (up to 1 year)
  Measured in blood, fasting
Metabolomics | Throughout the study (up to 1 year)
  Measured in blood and urin, fasting
Microbiomics | Throughout the study (up to 1 year)
  Measured in feces

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus N, Danmark, Denmark